CLINICAL TRIAL: NCT07349914
Title: An Investigation of Shoulder Pain and Function in Individuals With Implantable Cardiac Electronic Devices: A Prospective Study
Brief Title: Shoulder Pain and Function in Individuals With Implantable Cardiac Electronic Devices
Status: Enrolling by invitation | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, PT, PhD, Assoc. Prof., Hacettepe University
Other Study IDs: FTREK25/129
Record Dates: First submitted 2025-11-19; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Implantable Cardiac Electronic Devices; Pain; Upper Extremity; Posture; Function; Daily Activities
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with implantable cardiac electronic devices: Those who have recently undergone implantable cardiac electronic devices implantation Those scheduled for implantable cardiac electronic devices implantation Individuals with implantable cardiac electronic devices
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — Not applicable- observational study

SUMMARY:
The primary aim of our study is to evaluate shoulder pain, range of motion, postural changes, muscle tightness, activities of daily living, upper extremity functional status, and exercise capacity in individuals with Implantable Cardiac Electronic Devices (ICED), during each follow-up visit over a two-year period, and to compare the assessment outcomes according to different types of implantable cardiac electronic devices. The secondary aim of our study is to investigate the factors determining the severity and duration of shoulder pain in these patients.

DETAILED DESCRIPTION:
Implantable cardiac electronic devices have revolutionized the treatment of cardiac arrhythmias and significantly reduced the incidence of sudden cardiac death. The number of individuals living with these devices has increased substantially worldwide. Among implantable cardiac electronic devices are pacemakers, cardiac resynchronization therapy pacemakers or biventricular pacemakers, cardiac resynchronization therapy defibrillators, and implantable cardioverter defibrillators . Although cardiac device implantation is considered a minor surgical procedure, several complications may occur, including pocket hematoma, pneumothorax, wound infection, lead dislodgement, fracture, or perforation. In addition to these complications, it is well known that implantation may result in impaired ipsilateral upper extremity function, pain, and restricted shoulder range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older,
* Having an implantable cardiac electronic device
* Meeting the clinical indication for CIED implantation
* Without any complications at the most recent follow-up,
* Clinically stable for at least the past month, with any comorbid chronic conditions (e.g., hypertension, diabetes) well-controlled, considered suitable for assessment, and willing to provide informed consent to participate in the study.

Exclusion Criteria:

* Individuals with neurological, orthopedic, or psychiatric disorders,
* Individuals with a history of shoulder surgery or shoulder injury,
* Individuals with cognitive or mental impairments preventing comprehension of the study procedures, or those unwilling to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adults aged 18 years and older who have an implantable cardiac electronic device, including pacemakers, cardiac resynchronization therapy devices (CRT-P or CRT-D), or implantable cardioverter defibrillators (ICD).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-07-14 (Estimated); Study Completion 2027-08-14 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability | Follow-up over 2 years, with assessments every 6 months
  The Shoulder Pain and Disability Index (SPADI) will be used for assessment. The pain subscale comprises 5 items, and participants are asked to rate their pain over the past week during various movements using a Visual Analog Scale between 0 to 10 points. The disability subscale includes 8 items, assessing the level of difficulty experienced during different activities over the past week, also rated on a VAS from 0 (no difficulty) to 10 (unable to perform). Higher scores indicate greater pain and functional limitation. When the entire questionnaire is evaluated, a total score of 0 represents maximum well-being, whereas 130 represents the worst possible condition.
Assessment of Shoulder Range of Motion | Follow-up over 2 years, with assessments every 6 months
  A universal goniometer will be used to assess the range of motion of the shoulder. Active shoulder flexion, abduction, internal rotation, and external rotation will be measured in accordance with standard assessment principles. Each movement will be measured three times, and the average value will be recorded in degrees.
Assessment of Upper Extremity Functional Exercise Capacity | Follow-up over 2 years, with assessments every 6 months
  Unsupported Upper Limb Exercise Test (UULEX):Participants will be seated on a chair with their knees touching the wall where the UULEX lines are displayed. The UULEX consists of 8 horizontal levels, each 84 cm in width and 8 cm in height, with 15 cm between the centers of each level. The lowest line corresponds to the participant's knee level. Participants hold a plastic bar weighing 0.2 kg at shoulder width and move it from the hips toward the different levels of the UULEX lines. Each movement starts and ends at the hip joint. The first level is performed for 2 min, and each subsequent level is performed for 1 min. Using a metronome, participants lift the bar 30 times per min. Once participants reach their max height, the 0.2 kg bar is replaced with a 0.5 kg bar, and participants continue lifting to max height. Subsequently, the weight is increased by 0.5 kg per min at the specified level, up to max of 2 kg. Participants are instructed to continue the test until symptom limitation.
Tightness of muscle | Follow-up over 2 years, with assessments every 6 months
  Pectoralis minor and pectoralis major muscle tightness tests will be performed during musculoskeletal examination using a tape.

SECONDARY OUTCOMES:
Posture | Follow-up over 2 years, with assessments every 6 months
  Posture will be examined via the Corbin Postural Assessment Scale. The total points of the Corbin Postural Assessment Scale range from 0 to 28 points. A higher point represents worse posture.
Assessment of Musculoskeletal Pain | Follow-up over 2 years, with assessments every 6 months
  Musculoskeletal pain will be assessed using the Nordic Musculoskeletal Questionnaire (NMQ). This questionnaire evaluates symptoms (pain, discomfort, numbness) over the past 12 months in nine anatomical regions: neck, shoulders, elbows, wrists/hands, upper back, lower back, hips/thighs, knees, and ankles/feet. Participants are asked whether these symptoms have interfered with their work (at home or outside) during the past 12 months and whether they have experienced pain in any of these nine regions at any time during the past seven days.
Assessment of Upper Extremity Functional Status | Follow-up over 2 years, with assessments every 6 months
  Upper extremity functional status will be evaluated using the Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH) questionnaire. The QuickDASH is a shortened version of the full Disabilities of the Arm, Shoulder, and Hand questionnaire, consisting of 11 items. The scoring system is the same as the long version, using a 5-point Likert scale. According to this scale, upper extremity activity is rated as follows: 1 - no difficulty, 2 - mild difficulty, 3 - moderate difficulty, 4 - severe difficulty, and 5 - unable to perform. The total score ranges from 0 to 100, where 0 indicates no functional impairment and 100 indicates maximum functional limitation.
Assessment of Activities of Daily Living | Follow-up over 2 years, with assessments every 6 months
  The Nottingham Extended Activities of Daily Living Scale (NEADLS) will be used to evaluate participants' daily living activities across four subdomains: mobility, kitchen, domestic, and leisure activities. Responses are scored as follows: 0 = unable to perform, 1 = able to perform with assistance, 2 = able to perform independently but with difficulty, and 3 = able to perform independently and easily. The total score ranges from 0 to 66, with higher scores indicating greater independence in daily living activities.
Assessment of Body Awareness | Follow-up over 2 years, with assessments every 6 months
  Body awareness will be evaluated using the Body Awareness Rating Questionnaire. This questionnaire was developed to assess individuals' difficulties in perceiving and describing their bodily sensations and functions. It evaluates body awareness across four parameters: function, sensations, mood, and awareness. Each item is scored on a 7-point Likert scale. Each parameter receives a score ranging from 6 to 42, with higher scores indicating greater body awareness. Participants will be asked to read each statement within every parameter and select the score that best represents their experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Samanpazari, Turkey (Türkiye)